CLINICAL TRIAL: NCT07205198
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SIBP-A10 Injection in the Treatment of Advanced Malignant Tumor Subjects
Brief Title: A Clinical Trial of SIBP-A10 Injection in the Treatment of Advanced Malignant Tumor Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-A10-I
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Tumors
Keywords: Advanced malignant tumor; SIBP-A10; safety; efficacy; pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This study is an open-label, dose escalation, dose expansion, and indication expansion study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The subjects enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: SIBP-A10

INTERVENTIONS:
Drug: SIBP-A10 — SIBP-A10 injection. Strength: 0.5, 1.5, 3, 5, 7, 10 and 15 mg/kg. Intravenous infusion administration, with a treatment cycle of every 21 days, administered once on the first day of each cycle. The dose escalation stage,0.5 mg/kg group was subjected to accelerated titration, where the safety was evaluated within 21 days after the first administration to one subject. If unacceptable toxic reactions occurred, the traditional "3+3" dose escalation method was immediately switched. If unacceptable toxic reactions do not occur, the next dose group will be explored. The third stage will use RP2D for further exploration.

SUMMARY:
To evaluate the safety, tolerability of SIBP-A10 and determine the maximum tolerable dose (MTD) and phase II recommended dose (RP2D).

DETAILED DESCRIPTION:
This study is an open label, dose escalation, dose expansion, and indication expansion study to evaluate safety, tolerability, pharmacokinetics, preliminary anti-tumor efficacy, immunogenicity, impact on QT/QTc interval, and explore potential biomarkers of SIBP-A10 for injection in subjects with advanced metastatic tumors.

This study is divided into three stages and is planned to be set up seven dose groups, including 0.5, 1.5, 3, 5, 7, 10 and 15 mg/kg. The first stage is the dose escalation stage, which will start from the first and second doses for enrollment. If necessary, a 3+3 dose escalation design will be used. At least 19 subjects will be enrolled, and the specific sample size should be adjusted according to the subjects' tolerance level. The second stage is the dose expansion stage, where two or more doses are selected to enter the dose expansion phase, and at least 20 subjects will be enrolled in each dose group for dose expansion. The third stage is the indication expansion stage, where phase II recommended dose (RP2D) is preliminarily determined based on the escalation and expansion of dosage in the early stage. Using RP2D for indication expansion, we plan to expand four indication cohorts, with at least 40 subjects selected for each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study and sign an informed consent form;
* Age range of 18 to 75 years old (including boundary values), gender not limited;
* The clinical diagnosis of enrolled subjects should meet the conditions specified in the protocol:
* There must be at least one measurable lesion as the target lesion;
* Backfilling queue during dose escalation stage, dose expansion stage, and indication expansion stage: able to provide tumor tissue samples that meet the requirements of the protocol or undergo tumor biopsy during screening, or provide testing reports issued by legitimate testing institutions that meet the requirements;
* I have not received any medication targeting Siglec-15 in the past;
* The Eastern Cooperative Oncology Group (ECOG) physical fitness score ranges from 0 to 1;
* Expected survival period ≥ 3 months;
* During the screening period, the main organ functions were basically normal;
* During the screening period, women of childbearing age had negative blood pregnancy tests, and reproductive age subjects (including male subjects) had no pregnancy plans during the trial period and within 6 months after the last dose, and voluntarily took effective contraceptive measures.

Exclusion Criteria:

* The subject has the following tumors:

  * The subject has had other malignant tumors that have not healed within the past 5 years;
  * Subjects with meningeal metastases;
  * Subjects with active brain metastases;
* For anti-tumor subjects with a history of past treatment or surgery that does not comply with the protocol, or who have received treatment that does not comply with the protocol during the planned trial period
* Previous medical history or laboratory non-compliance with protocol requirements
* According to the researchers' assessment, the screening period is accompanied by severe, progressive, or uncontrolled non-tumor diseases, and it has been determined by the researchers that participating in the study would increase the risk for the subjects.
* According to the investigator's judgment, there are concomitant diseases (including but not limited to hypertension, diabetes, active infection, etc. that cannot be controlled by drugs) that seriously endanger the patient's safety or affect the patient's completion of the study
* Researchers determine that there are uncontrollable ascites, pleural effusion, or pericardial effusion, or those who have undergone ≥ 2 serosal drainage within 2 weeks prior to the first administration;
* Before starting treatment, the patient has not yet recovered to ≤ grade 1 from the toxic effects of previous treatments (including previous immunotherapy) and/or complications of previous surgical interventions.
* Individuals with a history of severe allergies to protein products, CHO cell products, other recombinant human or humanized antibodies, or components of the investigational drug;
* Pregnant and lactating women;
* Researchers believe that subjects who are not suitable to participate in this clinical study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
AE (Adverse Events) | From day 1 after the first dose to day 28 after the last dose
  That is adverse events, any adverse events that occurred to the subject during the study period.
Phase II recommended dose (RP2D) | Day 21 after the last dose in the dose expansion phase
  RP2D refers to the recommended dose determined through initial dose escalation and toxicity assessment in clinical trials, used for further evaluation of drug efficacy and safety.
Dose-limiting toxicity (DLT) | Day 21 after each dose in the dose escalation stage
  DLT is defined as any adverse event related to the drug defined in the protocol that occurs within 21 days of the first cycle after a single administration.
Maximum tolerated dose (MTD) | Day 21 after the last dose in the dose escalation stage
  MTD is defined as the maximum dose at which the number of DLT cases occurring during the DLT observation period within 21 days after a single administration is ≤ 1/6 of the total number of cases.

SECONDARY OUTCOMES:
AUC (Area Under The Plasma Concentration Versus Time Curve) | Day 1, Day 22 and Day 64 after the first dose
  It shows the degree to which a drug is absorbed and used in the body.
Cmax (Peak Plasma Concentration) | Day 1, Day 22 and Day 64 after the first dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax (Peak Time) | Day 1, Day 22 and Day 64 after the first dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the subject plasma concentration curve after administration.
ORR (Objective Response Rate) | 6 weeks after the last evaluation
  The proportion of subjects whose tumor volume shrinks to a predetermined value and maintains the minimum time limit and is the sum of complete and partial responses.
DCR (Disease control rate) | 6 weeks after the last evaluation
  In clinical trials, the percentage of subjects with advanced cancer who responded fully to cancer treatment, partially responded, and had stable disease.
PFS (Progression-free survival) | 6 weeks after the last evaluation
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
OS (overall survival) | From the first injection to 36 months after the first injection.
  From randomization to time of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Docter, Principal Investigator — Shanghai Institute Of Biological Products
Locations (1):
- Zhongshan Hospital Affiliated to Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No